CLINICAL TRIAL: NCT02746081
Title: An Open-label, Non-randomized, Multicenter Phase I Study to Determine the Maximum Tolerated or Recommended Phase II Dose of Oral Mutant IDH1 Inhibitor BAY1436032 and to Characterize Its Safety, Tolerability, Pharmacokinetics and Preliminary Pharmacodynamic and Anti-tumor Activity in Patients With IDH1-R132X-mutant Advanced Solid Tumors
Brief Title: Phase I Study of BAY1436032 in IDH1-mutant Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18239; 2015-003483-37 (EudraCT Number)
Record Dates: First submitted 2016-04-08; First posted 2016-04-21 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumors
Keywords: BAY1436032; Solid tumors; IDH1; Cancer; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Efficacy; Food-effect
MeSH Terms: conditions — Neoplasms | interventions — BAY 1436032

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY1436032 (Experimental): Dose escalation: Patients with any type of IDH1-R132X-mutant solid tumor may be eligible for enrollment. A minimum of 3 patients per cohort will be treated. If dose limiting toxicities (DLTs) occur, Bayesian dose-DLT modeling will be performed to help guide dosing decisions and to identify the maximum tolerated dose (MTD). If the MTD is not reached, a recommended phase II dose (RP2D) will be chosen based on available safety, tolerability, PK, PD and clinical efficacy data.
  Dose expansion: The dose and schedule that was determined to be most appropriate in the dose escalation part of the study, which may be the MTD and / or the RP2D, will be used. Cohorts will consist of patients with the following IDH-R132X-mutant tumor types: (1) anaplastic glioma; (2) glioblastoma; (3) intrahepatic cholangiocarcinoma; (4) tumor types other than those in Cohorts 1-3.
  Interventions: Drug: BAY1436032

INTERVENTIONS:
Drug: BAY1436032 — The selected starting dose of BAY1436032 is 300 mg/day (150 mg BID) to be administered orally continuously in tablet form in 21-day cycles. Adjustments to this schedule may be made if warranted by information collected during the course of the study. The maximum feasible dose of BAY1436032 is expected to be 3000 mg/day.

SUMMARY:
The primary objective of this study is:

- Determine the safety, tolerability, maximum tolerated dose (MTD) or recommended Phase II dose (RP2D) of BAY 1436032 in patients with isocitrate dehydrogenase-1 (IDH1)-R132X-mutant advanced solid tumors.

The secondary objectives of this study are:

* Evaluate the pharmacokinetics (PK) of BAY1436032 in patients with IDH1-R132X-mutant advanced solid tumors.
* Evaluate the effect of a standard high-fat, high calorie meal on the PK of BAY1436032.
* Assess pharmacodynamic (PD) effects and evidence of clinical efficacy associated with BAY1436032 administration in patients with IDH1-R132X-mutant advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Patients with a histologically confirmed solid tumor:

  * Tumor must harbor an IDH1-R132X mutation
  * Disease must be evaluable as per RECIST 1.1 or RANO (for gliomas). At least one measurable target lesion is required in expansion cohort patients
  * Patients with advanced cancer who are refractory to, have demonstrated intolerance to, or have refused access to, available standard therapies
  * Glioma patients must have completed chemoradiotherapy at least 12 weeks prior to screening and their baseline scan
* Patient must be able to provide a formalin-fixed and paraffin-embedded (FFPE) tumor tissue specimen prior to treatment. The specimen may have been taken at any time during the course of the disease and may be from the primary tumor or from a metastasis
* Patient must be able to take oral medication and comply with protocol procedures and scheduled visits
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Negative serum or urine pregnancy test must be obtained within 7 days prior to the first dose of study drug in women of childbearing potential. Negative results must be available prior to study drug administration. Pregnancy tests will be repeated regularly during treatment
* Sexually active women and men of reproductive potential must agree to use highly effective contraception. This applies for the period between signing of the informed consent and 3 months after the last administration of study drug. These procedures should be documented in source documents. The investigator or a designated associate is requested to advise the patient on how to achieve highly effective birth control. Highly effective contraception includes:

  * Established use of oral, injected or implanted hormonal methods of contraception
  * Placement of certain intrauterine devices (IUD) or intrauterine systems (IUS)
  * Hysterectomy, or vasectomy of the partner (provided that partner is the sole sexual partner of the woman of childbearing potential trial participant and that the vasectomized partner has received medical assessment of the surgical success) In addition, the use of condoms for patients or their partners is required
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent, including consent for biomarker analyses, must be obtained prior to any study-specific procedures
* Adequate blood clotting as defined by international normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN (patients on anticoagulation with an agent such as warfarin or heparin or rivoraxaban will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists). For patients on warfarin, close monitoring of at least weekly evaluations will be performed until INR is stable based on a measurement at pre-dose, as defined by the local standard of care
* Adequate bone marrow, liver, and renal functions as assessed by the following laboratory requirements to be conducted within 7 days prior to the first dose of study drug:

  * Hemoglobin ≥ 9.0 g/dL;
  * Absolute neutrophil count (ANC) ≥ 1.5x10^9/L;
  * Platelet count ≥ 100x10^9/L.
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN). For intrahepatic cholangiocarcinoma (IHCC) patients only, total bilirubin ≤ 2.5 times ULN is acceptable
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN (≤ 5 times ULN for patients with impaired liver function due primary tumor or metastatic disease)
  * Estimated glomerular filtration rate (eGFR) ≥ 40 mL/min per 1.73 m^2 according to the Modification of Diet in Renal Disease Study Group (MDRD) formula
* Minimum life expectancy of 3 months per the judgment of the investigator

Exclusion Criteria:

* Known hypersensitivity to the study drug or excipients of the preparation or any agent given in association with this study
* History of cardiac disease, including congestive heart failure of New York Heart Association (NYHA) class >II, unstable angina (anginal symptoms at rest) or new-onset angina (within 6 months prior to study entry), myocardial infarction within 6 months prior to study entry, or cardiac arrhythmias requiring anti-arrhythmic therapy except for beta-blockers and digoxin; evidence for uncontrolled coronary artery disease (e.g. angina pectoris, myocardial infarction within 6 months prior to study entry, major regional wall motion abnormalities upon baseline echocardiography or multiple-gated acquisition [MUGA] scan). Patients with a pacemaker are also excluded
* Left ventricular ejection fraction (LVEF) < 40% as measured by echocardiography or MUGA scan performed at Screening
* Uncontrolled hypertension defined as systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg, despite medical management
* Patients who have an active clinically significant infection of the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 2
* Previous or coexisting cancer(s) distinct in primary site or histology from the cancer evaluated in this study EXCEPT:

  * Appropriately treated cervical cancer in-situ, non-melanoma skin cancers, or superficial bladder tumors (Ta and Tis)
  * Any cancer that was curatively treated at least 3 years before entry into this study
* Unresolved specific chronic toxicity of previous treatment of grade > 1 except for alopecia or hemoglobin ≤9.0 g/dL (or ≤5.6 mmol/L)
* Major surgery, significant trauma, wide-field radiotherapy, or therapy with monoclonal antibodies within 4 weeks before the first dose of study drug
* Treatment with investigational or approved anti-cancer drugs within 4 weeks before the start of BAY1436032 treatment and during the study (glioma patients must have completed chemoradiotherapy at least 12 weeks prior to screening and their baseline scan; see inclusion criteria #2)
* Pregnant women. Women of reproductive potential must have a negative serum or urine pregnancy test performed within 7 day
* Prior treatment with any therapy targeting mutant IDH1 (including BAY1436032)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of BAY1436032 | 21 days
  MTD is defined as the maximum dose at which the predicted incidence of DLTs during Cycle 1 (DLT evaluation period) is ≤25%.
Number of participants with adverse events as a measure of safety and tolerability of BAY1436032 | Up to 30 months
  Safety and tolerability variables will include AEs, laboratory safety tests, ECGs, and vital signs.
Recommended Phase II Dose (RP2D) of BAY1436032 | Up to 20 months
  If the MTD is not reached, the primary variable will be the RP2D, defined based on all available safety, PK, PD, biomarker, and efficacy data collected after the start of BAY1436032 treatment.

SECONDARY OUTCOMES:
Objective response rate (partial and complete response) | Up to 30 months
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or for gliomas Response Assessment in Neuro-Oncology (RANO)
Duration of response | Up to 30 months
Progression free survival (PFS) | Up to 30 months
  For expansion part only
Cmax of BAY1436032 | on C1D-2 and C1D1
AUC(0-12) of BAY1436032 | on C1D-2 and C1D1
AUC(0-24) of BAY1436032 | on C1D-2 and C1D1
C(max,md) of BAY1436032 | on C1D15
AUC(0-12)md of BAY1436032 | on C1D15
Change of 2-hydroxyglutarate (2-HG) concentration in plasma from baseline | Up to 30 months
Change of 2-hydroxyglutarate (2-HG) concentration in urine from baseline | Up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- United States (3):
  - Los Angeles, California
  - Houston, Texas
  - Charlottesville, Virginia
- København Ø, Denmark
- Germany (5):
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Essen, North Rhine-Westphalia
- Japan (3):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Chuo-ku, Tokyo